CLINICAL TRIAL: NCT06069583
Title: Using the Support Online Platform for Self-management Education of Adults Living With Type 1 Diabetes as Part of Usual Care or Independently: an Implementation Study
Brief Title: Implementation of Support in the Care of Adults Living With Type 1 Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: Institut de Recherches Cliniques de Montreal (Other); Centre Hospitalier de l'Universite Laval (CHUL) (Unknown); Centre hospitalier de l'Université de Montréal (CHUM) (Other); Centre de médecine métabolique de Lanaudière (Unknown)
Responsible Party: Principal Investigator, Anne-Sophie Brazeau, Associate Professor, McGill University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MP-02-2024-11714
Record Dates: First submitted 2023-09-29; First posted 2023-10-06 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Type 1 Diabetes; Metabolic Disease; Endocrine System Diseases; Autoimmune Diseases; Immune System Diseases
Keywords: self-management education; Hemaglobin A1c; Online education; adults; type 1 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Metabolic Diseases; Endocrine System Diseases; Autoimmune Diseases; Immune System Diseases

STUDY DESIGN:
Intervention Model Description: mixed-method multi-site, 2 arms, non-randomized, type 1 hybrid effectiveness-implementation trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Support integrated in usual care (Experimental): PWT1D participants will have access to Support as part of their regular care (their HCPs will use Support in their care). PWT1D participants in ARM 1 are followed in one of the 4 participating clinics either in-person or remotely or hybrid.
  Interventions: Behavioral: Support platform
- Support through independent access (Active Comparator): PWT1D participants will have access to Support, independently from their regular care (they may initiate discussion about the platform with their diabetes care team who might register themselves on the platform, but will not prompt to any specific section on the platform and will not receive any training about the platform). PWT1D participants in ARM 2 can be followed in any other clinics in Canada.
  Interventions: Behavioral: Support platform

INTERVENTIONS:
Behavioral: Support platform — The study will be conducted over a 12-month period. This should allow participants to see their medical team 2 to 3 times during this timeframe. Participants of arms 1 and 2 will have access to the Support platform and will receive a monthly newsletter, informing them of news on the platform and acting as a reminder to log in. Several features are included in this responsive-designed platform to enhance participation, such as a visual of personal progress, ability to bookmark content, change their avatar.
  Support contains 3 main components: Educational material, News blog written by HCPs weekly in collaboration with patient-partners on up-to-date topics related to T1D, a peer-to-peer discussion forum which is moderated daily by a HCP specializing in T1D.

SUMMARY:
The investigators will conduct a trial to evaluate if an online training and support platform can help adults living with type 1 diabetes (T1D) in their diabetes self-management. Investigators will compare a group that has access to the "Support" platform through their usual medical care to a group that accesses the platform independently. The first group will be recruited through four participating clinics in the province of Quebec (Canada). The second group will be composed of adults living with T1D across Canada. Participants will have access to the platform for 12 months and will be asked to complete online questionnaires at the beginning and after 6 and 12 months, and share their glucose reader data with the research team. A subgroup of participants as well as healthcare professionals from the four clinics will be invited to participate in an individual interview aiming to understand the barriers and facilitators of integration "Support" in clinical care.

DETAILED DESCRIPTION:
Type 1 diabetes (T1D) is a chronic condition which requires life-sustaining insulin therapy as well as knowledge, skills and confidence to self-manage. Tailored diabetes self-management education (DSME) should be offered to all people living with diabetes (PWT1D) at diagnosis, but also in a timely manner according to needs. DSME has the potential to improve quality of life and decrease diabetes complications. Despite the positive outcomes of other DSME programs, participation rates of DSME vary greatly perhaps because access remains sub-optimal. Also, healthcare professionals (HCPs) face a challenge to remain aware of the particularities of T1D and stay up-to-date on the rapidly evolving evidence-based knowledge, technologies and therapies available. The investigators propose to examine an online training and peer support platform, called "Support" as a potential alternative for DSME.

The overall purpose of this hybrid effectiveness-implementation study is to investigate if integrating the "Support" platform to routine medical care of adults living with T1D (i.e., diabetes team referring to the "Support" platform during appointments) can improve diabetes self- management, in comparison with navigating the "Support" platform independently of usual care (i.e., the platform not being discussed during appointment) (Effectiveness), and to study the factors affecting its implementation in real-life settings (Implementation).

This study is a mixed-method multi-site, 2 arms, non-randomized, type 1 hybrid effectiveness-implementation trial.

ARM 1: PWT1D participants will have access to Support as part of their regular care (their HCPs will use "Support" in their care). PWT1D participants in ARM 1 are followed in one of the 4 participating clinics either in-person or remotely or hybrid.

ARM 2: PWT1D participants will have access to "Support", independently from their regular care (they may initiate discussion about the platform with their diabetes care team who might register themselves on the platform, but will not prompt to any specific section on the platform and will not receive any training about the platform). PWT1D participants in ARM 2 can be followed in any other clinics in Canada.

Implementation data will be gathered through HCP participants in the participating clinics.

Participants will have to answer online surveys at baseline, 6 months and 12 months. After completing the baseline questionnaire, they will receive an access to the platform. A subgroup of participants as well as participating HCPs will be invited for individual interviews to discuss their experience in using the platform.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of T1D (including LADA - latent autoimmune diabetes in adults)
* Have access to Internet
* Use of an active email address
* Comprehension of English or French
* Live in Canada

Exclusion Criteria:

- Unable to use the Support platform

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322 (Estimated)
Dates: Start 2024-05-05 (Actual); Primary Completion 2027-05-05 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Self-efficacy for diabetes management | 0, 6 and 12 months
  Diabetes Self-Management Questionnaire-Revised (DSMQ-R; 27-items, score on 10)

SECONDARY OUTCOMES:
Well-being | 0, 6 and 12 months
  WHO-5 well-being index
Continuous Glucose Monitoring (CGM) - % Time in range | 0, 6 and 12 months
  % Time in range (3.9-10.0mmol/L) over the past 4 weeks. Participants may share their account access so the research team will be able to export data or may upload a PDF of their data through REDCap.
Continuous Glucose Monitoring (CGM) - % Time above range | 0, 6 and 12 months
  % Time above range (3.9-10.0mmol/L) over the past 4 weeks. Participants may share their account access so the research team will be able to export data or may upload a PDF of their data through REDCap.
Continuous Glucose Monitoring (CGM) - % Time below range | 0, 6 and 12 months
  % Time below range (3.9-10.0mmol/L) over the past 4 weeks. Participants may share their account access so the research team will be able to export data or may upload a PDF of their data through REDCap.
Continuous Glucose Monitoring (CGM) - Standard deviation | 0, 6 and 12 months
  Standard deviation of the past 4 weeks. Participants may share their account access so the research team will be able to export data or may upload a PDF of their data through REDCap.
Continuous Glucose Monitoring (CGM) - % Coefficient of variation | 0, 6 and 12 months
  % Coefficient of variation of the past 4 weeks. Participants may share their account access so the research team will be able to export data or may upload a PDF of their data through REDCap.
Hemoglobin A1c | 0, 6 and 12 months
  self-reported last Hemoglobin A1c (date and value) through online questionnaire
Severe hypoglycemic events | 0, 6 and 12 months
  Self-reported severe hypoglycemic events in the past 6 months
Diabetic Ketoacidosis (DKA) events | 0, 6 and 12 months
  Self-reported DKA events in the past 6 months
calls to 911 | 0, 6 and 12 months
  Self-reported number of calls to 911 in the past 6 months
calls to 811 | 0, 6 and 12 months
  Self-reported number of calls to 811 in the past 6 months
Cost effectiveness (self-efficacy) | 6 and 12 months
  Cost effectiveness of access to Support as part of usual care compared with independent access in terms of incremental cost effectiveness ratio (ICER) for self-efficacy
Cost effectiveness (HbA1c) | 6 and 12 months
  Cost effectiveness of access to Support as part of usual care compared with independent access in terms of incremental cost effectiveness ratio (ICER) for HbA1c

OTHER OUTCOMES:
Implementation question | 0 month
  Participants will be asked where they heard about the platform.
communication with health care team | 0, 6 and 12 months
  Question about type (in-person, phone, video call or email) and frequency of communication with health care team
Engagement with Support platform (T1D patient) - time in minutes on platform | 6, 12 months
  Engagement metrics will be extracted using Google analytics - time (minutes) spent on the platform
Engagement with Support platform (T1D patient) - total pages viewed | 6, 12 months
  Engagement metrics will be extracted using Google analytics - total pages viewed from the platform
Engagement with Support platform (T1D patient) - downloaded documents | 6, 12 months
  Engagement metrics will be extracted using Google analytics - downloaded documents from the platform
Engagement with Support platform (T1D patient) - use of calculators | 6, 12 months
  Engagement metrics will be extracted using Google analytics - use of calculators on the platform
Engagement with Support platform (Health Care Provider) - time in minutes on platform | 6, 12 months
  Engagement metrics will be extracted using Google analytics - time (minutes) spent on the platform
Engagement with Support platform (Health Care Provider) - content accessed | 6, 12 months
  Engagement metrics will be extracted using Google analytics - specific content accessed from the platform
Engagement with Support platform (Health Care Provider) - total pages viewed | 6, 12 months
  Engagement metrics will be extracted using Google analytics - total pages viewed from the platform
Engagement with Support platform (Health Care Provider) - downloaded documents | 6, 12 months
  Engagement metrics will be extracted using Google analytics - downloaded documents from the platform
Engagement with Support platform (Health Care Provider) - use of calculators | 6, 12 months
  Engagement metrics will be extracted using Google analytics - use of calculators on the platform
Satisfaction with Support-t platform - T1D patient | 6, 12 months
  Satisfaction will be rated on a scale from 1 to 10. Higher scores indicate greater satisfaction with the platform.
Experience with Support platform (Barriers, facilitators, satisfaction, fidelity) - T1D patient | 12 months
  Individual interviews to understand the experience in the context of implementation of the Support-t platform (Barriers, facilitators, satisfaction, fidelity) using qualitative descriptive methodology
Experience with Support platform (Barriers, facilitators, satisfaction, fidelity) - Health Care Provider | 12 months
  Individual interviews to understand the experience in the context of implementation of the Support-t platform (Barriers, facilitators, satisfaction, fidelity) using qualitative descriptive methodology

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Sophie Brazeau, PhD, Principal Investigator — School of human nutrition - McGill University
Locations (4):
- Canada (4):
  - Institut de recherches cliniques de Montréal, Montreal, Quebec
  - Centre hospitalier de l'université de Montreal, Montreal, Quebec
  - Centre hospitalier de Quebec, Université Laval, Québec, Quebec
  - Centre de médecine métabolique de Lanaudière, Terrebonne, Quebec

REFERENCES:
- [Background] Xie LF, Roy-Fleming A, Haag S, Costa DD, Brazeau AS. Development of the Support self-guided, web application for adults living with type 1 diabetes in Canada by a multi-disciplinary team using a people-oriented approach based on the Behaviour Change Wheel. Digit Health. 2023 Jan 24;9:20552076231152760. doi: 10.1177/20552076231152760. eCollection 2023 Jan-Dec. PMID 36762025
- [Background] Xie LF, Itzkovitz A, Roy-Fleming A, Da Costa D, Brazeau AS. Understanding Self-Guided Web-Based Educational Interventions for Patients With Chronic Health Conditions: Systematic Review of Intervention Features and Adherence. J Med Internet Res. 2020 Aug 13;22(8):e18355. doi: 10.2196/18355. PMID 32788152
- [Background] Kruger J, Brennan A, Thokala P, Basarir H, Jacques R, Elliott J, Heller S, Speight J. The cost-effectiveness of the Dose Adjustment for Normal Eating (DAFNE) structured education programme: an update using the Sheffield Type 1 Diabetes Policy Model. Diabet Med. 2013 Oct;30(10):1236-44. doi: 10.1111/dme.12270. Epub 2013 Aug 19. PMID 23815547
- [Background] Stanton-Fay SH, Hamilton K, Chadwick PM, Lorencatto F, Gianfrancesco C, de Zoysa N, Coates E, Cooke D, McBain H, Heller SR, Michie S; DAFNEplus study group. The DAFNEplus programme for sustained type 1 diabetes self management: Intervention development using the Behaviour Change Wheel. Diabet Med. 2021 May;38(5):e14548. doi: 10.1111/dme.14548. Epub 2021 Mar 10. PMID 33617669
- [Background] Pereira K, Phillips B, Johnson C, Vorderstrasse A. Internet delivered diabetes self-management education: a review. Diabetes Technol Ther. 2015 Jan;17(1):55-63. doi: 10.1089/dia.2014.0155. PMID 25238257
- [Background] Curran GM, Bauer M, Mittman B, Pyne JM, Stetler C. Effectiveness-implementation hybrid designs: combining elements of clinical effectiveness and implementation research to enhance public health impact. Med Care. 2012 Mar;50(3):217-26. doi: 10.1097/MLR.0b013e3182408812. PMID 22310560
- [Background] Schmitt A, Kulzer B, Ehrmann D, Haak T, Hermanns N. A Self-Report Measure of Diabetes Self-Management for Type 1 and Type 2 Diabetes: The Diabetes Self-Management Questionnaire-Revised (DSMQ-R) - Clinimetric Evidence From Five Studies. Front Clin Diabetes Healthc. 2022 Jan 13;2:823046. doi: 10.3389/fcdhc.2021.823046. eCollection 2021. PMID 36994332